CLINICAL TRIAL: NCT06854614
Title: Sequential or CombinaTion Anti-obesitY Medication With Muscle Preservation for Weight Loss and MaintEnance: A PragmAtic Randomized CoNtrolled Trial (STAY-LEAN Trial)
Acronym: STAY-LEAN
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Bartolome Burguera, Institute Chief, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-695
Record Dates: First submitted 2025-02-21; First posted 2025-03-03 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Qsymia; Naltrexone-Bupropion combination; bupropion hydrochloride, naltrexone hydrochoride drug combination; Orlistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 AOM (Experimental): Comprehensive weight loss Program + Enhanced lifestyle changes + Group 1 AOM sequential therapy (phentermine-topiramate or naltrexone-bupropion)
  Interventions: Other: Comprehensive weight loss; Other: Enhanced lifestyle changes; Drug: Phentermine-Topiramate; Drug: Naltrexone-Bupropion Combination
- Group 2 AOM (Experimental): Comprehensive weight loss + Enhanced lifestyle changes + Group 2 AOM Sequential therapy (orlistat)
  Interventions: Other: Comprehensive weight loss; Other: Enhanced lifestyle changes; Drug: Orlistat

INTERVENTIONS:
Other: Comprehensive weight loss — Shared Medical Appointments
Other: Enhanced lifestyle changes — Subjects will also be referred to an exercise physiologist for a personalized physical activity program. Physical Activity and Exercise will be discussed during SMAs as well and individually as needed for exercise progression The participants exercise prescription will be individualized based on an initial assessment. Exercise duration and progression will be recommended at the discretion of staff and exercise physiologist. The exercise program will be structured but flexible, which means patients can substitute group exercises with individual exercise if necessary, following the FITT-VP format (frequency, intensity, time, type, volume and progression). Patients can reduce exercise frequency if the duration is prolonged, or intensity is increased. Investigators will encourage patients to use Cleveland Clinic gyms across the enterprise.
Drug: Phentermine-Topiramate — Medication for chronic weight management (Rx)
  Other Names: Qsymia
  Arms: Group 1 AOM
Drug: Naltrexone-Bupropion Combination — Medication for chronic weight management (Rx)
  Other Names: Contrave
  Arms: Group 1 AOM
Drug: Orlistat — Medication for chronic weight management (Rx)
  Other Names: Xenical
  Arms: Group 2 AOM

SUMMARY:
This is a prospective, pragmatic, 21 month, single-center, randomized, 2-phased, open-label, parallel-group trial comparing the use of enhanced lifestyle changes (ELC) in two different sequential anti obesity medication (AOM) therapies. The ELC consists of a medically-supervised and comprehensive weight loss program (Cleveland Clinic's Department of Endocrinology, Diabetes and Metabolism's Integrated Weight Management Program). In the first phase (9 months) of the study, all participants will receive tirzepatide 15 mg (option #1) or semaglutide 2.4 mg if tirzepatide is not tolerated. In the second phase, after completing 9 months of tirzpeatide or semaglutide, participants will continue ELC and will be randomly assigned to a different oral AOM therapy for another 12 months: group 1 (phentermine-topiramate or naltrexone-bupropion) or group 2 (orlistat).

The primary endpoint will be the percentage weight loss at 21 months compared to weight loss at 9 months. The goal will be to show superiority of the arm receiving ELC plus AOM therapy (phentermine-topiramate or naltrexone-bupropion) when compared to the other AOM therapy group (orlistat). Secondary and exploratory endpoints will include percentage of fat mass loss, lean muscle mass, functional capacity, muscle strength and compliance to enhanced lifestyle changes. Informed consent will be obtained. IRB approval of the study will be obtained.

DETAILED DESCRIPTION:
Obesity is the most prevalent disease and affects nearly 40% of adults in the US and it is a major risk factor for several chronic diseases including hypertension, dyslipidemia, T2D, depression, coronary heart disease, stroke, osteoarthritis, obstructive sleep apnea (OSA), fatty liver disease, and some cancers, to name a few. Patients with obesity have an increased risk of all-cause and cardiovascular death. In recognition of the biologic basis and seriousness of obesity, several professional health associations and organizations worldwide recognize obesity as a disease . Obesity is often stigmatized and viewed as a personal choice or lack of willpower, rather than a chronic disease, complex disease that can result from a combination of genetic, environmental, and behavioral factors, including diet and physical activity levels.

Obesity is one of the biggest drivers of preventable chronic diseases and healthcare costs in the United States. Currently, estimates for these costs are $497 billion per year in direct health care costs, and $1.24 trillion in indirect costs due to lost productivity in 2016. In addition, obesity is associated with job absenteeism and with lower productivity while at work costing approximately $4.3 billion annually.

Cleveland Clinic is one of the largest hospital systems in the United States, employing approximately 70,000 individuals, most of whom are enrolled in the Cleveland Clinic's Employee Health Plan for their medical insurance. Of the approximately 70,000 adult employees and their spouses on the Health Plan, approximately 22,000 have obesity, defined by BMI ≥ 30 kg/m2, and more than 8,000 suffer severe obesity (BMI ≥ 35 kg/m2). Cleveland Clinic's Employee Health Plan (EHP) provides employees diagnosed with obesity support for participating in a weight management program (part of our Healthy Choice program). Caregivers and their spouses who participate can improve their health and get up to 30% off their premiums by meeting personalized annual medical, nutrition or fitness goals. In 2022, only 40% of employees with obesity signed up for the Healthy Choice program.

In the US, employers are the ultimate purchasers of health care for the majority (56%) of employees. Recommendations support addressing obesity in the workplace; however, real-world evidence of best practices for chronic weight management in the employer context is still lacking. More specifically, the impact of aggressively managing obesity (i.e., the primary problem) including the use of anti-obesity medications (AOMs) is still poorly studied. In order for medications for chronic weight management to be included in the health care offered to employees, employers have to "opt-in" or deliberately decide to pay for these medications for employees, even when payers have added them to their formulary. Despite the potential benefits of these medications, the high cost may limit their accessibility and effectiveness in managing obesity. Recent studies still show that the use of anti-obesity medications are under prescribed, as only one percent of office-based visits for patients with obesity received a prescription for an AOM. More recently, the coverage of anti-obesity medications is expanding across the country, and many federal and state employers, including Medicaid in some states, are now covering AOM therapy.

AOMs are often required as adjuvant therapy for obesity in combination with lifestyle interventions, especially long-term to avoid weight regain. Weight plateau and regain is due to reduction of total energy expenditure due to lean and fat mass loss, in addition to increased appetite due to metabolic adaptation and is often seen once AOM therapy are stopped. Sustainable caloric restriction is not practical in the long-term due changes in metabolic adaptation, metabolic rate and lean muscle mass. Lifestyle interventions encouraging increased physical activity, some caloric restriction and AOMs are helpful for sustainable weight loss, highlighting the importance of developing effective strategies for weight loss maintenance beyond the initial weight loss. In addition to that, sequential pharmacotherapy has emerged as a promising approach for the treatment of obesity, especially for patients who have not achieved adequate weight loss with initial therapy. The use of multiple medications with different mechanism of action can enhance weight loss by targeting different pathways involving energy balance and appetite regulation. New weight management therapies are promising but costs can be prohibitive and long-term treatment sometimes is not feasible. Findings alternative strategies that can maintain the initial weight loss or avoid weight regain are needed. More research is needed to better understand the safety and efficacy of sequential therapy for the treatment of obesity, particularly for long-term weight loss maintenance. Obesity treatment should also go far beyond achieving weight loss: weight is only one measurement for obesity treatment. Preservation of muscle mass, aerobic fitness and body composition, which have cardiovascular and metabolic implications, are often benefits observed when exercise programs are incorporated into weight loss programs.

Our weight management group has extensive experience treating obesity and has developed novel approaches for obesity management. In one of our previous trials, the investigators found greater weight loss with an employer sponsored weight management program augmented with AOMs vs the weight management program (WMP) alone.24 The proposed trial will afford the opportunity to study the effects of a well-established weight management program based on a strong foundation of lifestyle intervention, leveraging a quality diet and focusing on muscle and strength preservation through exercise, augmented with AOM therapy to control appetite. The lifestyle intervention program in this trial will be administered through shared medical appointments SMAs (monthly for the first 13 months, every other month from month 13 to 21), which is a concept based on the chronic care model that combines group appointments for patients with clinical intervention, consisting of encounters with a nutritionist, exercise physiologist, and endocrinologist/obesity medicine specialist. The pharmacologic interventions under study will use FDA-approved medications for chronic weight management in a sequential fashion, approaches that have not been studied extensively.

Cleveland Clinic provides a unique environment to investigate the impact of a weight-centric program, including the utilization of approved medications for chronic weight management in patients with obesity, in the context of an employer-based weight management program. The use of a pragmatic clinical trial (PCT) design aims to study the effects of a weight management program that includes treatment with medication for chronic weight management in an employer-based real-world setting while employing a prospective comparison between two randomly assigned pharmacologic intervention strategies in employees with obesity.

The main objective of this randomized pragmatic clinical trial is to evaluate if switching patients (sequential therapy) from a highly effective (and more costly) AOM (GLP-1RA or GIP/GLP-1 dual agonist) to an oral (and cheaper) AOM leads to a significant and sustainable weight loss and to evaluate the importance of a weight management program focusing on a healthy diet and an exercise, with the goal of muscle mass preservation, can have additional benefits when combined with AOM.

ELIGIBILITY:
Inclusion Criteria:

1. Gender: men and women
2. Ethnicity: all ethnic groups
3. Age: ≥ 25, < 65 years

5. Obesity, BMI ≥ 30 and BMI < 45 6. An Employee, or the significant other of an employee, that is covered by the Cleveland Clinic Employee Health Plan

Exclusion Criteria:

1. Patients with history of diabetes
2. Glomerular Filtration Rate <30 mL/min/1.73 m2 (calculated by the Chronic Kidney Disease Epidemiology Collaboration Equation, CKD-EPI)
3. Current glucocorticoid therapy, except for maintenance glucocorticoid therapy of prednisone 5 mg or equivalent
4. Currently or within the past 6 months receiving an anti-obesity medication, or any other medication used for the primary intent of weight loss
5. Any condition, unwillingness, or inability, not covered by any of the other exclusion criteria, which, in the study clinician's opinion, might jeopardize the subject's safety or compliance with the protocol
6. Mental incapacity or language barrier
7. Pregnancy or plans to become pregnant within the next 2 years
8. Personal or family history of medullary thyroid carcinoma
9. Personal or family history of Multiple Endocrine Neoplasia syndrome type 2
10. previous history of pancreatitis, history of severe liver disease (Cirrhosis), or severe disease of digestive tract
11. History of congestive heart failure
12. History of bariatric or metabolic surgery/procedure
13. Prior participation in the Endocrinology and Metabolism Institutes Integrated Weight Management Program within the past 3 months
14. Contraindication for physical activity or significant physical limitation
15. Smoking
16. Cardiovascular disease including uncontrolled hypertension, history of arrhythmias or coronary artery disease
17. History of recurrent kidney stones
18. History of glaucoma
19. History of seizure disorders
20. Uncontrolled lung disease (difficult to control Asthma or COPD)
21. Medications that affect physical performance (beta-blocker or others)
22. Uncontrolled thyroid disease
23. Patients with personal commitments that limit optimal participation
24. Concurrent use of bupropion or naltrexone or previous intolerance to any of these medic
25. Previous intolerance to use or allergy to any of the anti-obesity medications approved in this study
26. History of malabsorptive disorders or cholestasis
27. Conductive implanted devices (i.e. cardiac pacemaker, cardioverter-defibrillators)

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-04-28 (Estimated); Study Completion 2028-04-28 (Estimated)

PRIMARY OUTCOMES:
Weight change | month 9 to month 21
  Weight change from month 9 month to month 21 in body weight (%) between both arms

SECONDARY OUTCOMES:
Change in body weight % | baseline to month 21
  Change from baseline to month 9, 15 and 21 in body weight (%)

CONTACTS AND LOCATIONS:
Overall Officials: Bartolome Burguera, M.D, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No